CLINICAL TRIAL: NCT06624449
Title: The Effect of Hot and Cold Debriefing on BLS Competence and Reflection In Undergraduate Nursing Students.
Brief Title: The Effect of Immediate Versus Delayed Debriefing on Basic Life Support Competence In Undergraduate Nursing Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Fahad Alanezi, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-0423
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: BLS Competence; Debriefing
Keywords: Debriefing; Simulation; Basic Life Support; Undergraduate Nursing Students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Debriefing (Experimental): The researcher assigned a cold debriefing (after one-day post-simulation) for undergraduate nursing students in the intervention group.
  Interventions: Behavioral: Cold debriefing
- Hot Debriefing (Other): The control group received a hot debriefing (immediately after the simulation).
  Interventions: Behavioral: Hot Debriefing

INTERVENTIONS:
Behavioral: Cold debriefing — Manipulation (experimental): The researcher assigned a cold debriefing (after one-day post-simulation) for undergraduate nursing students in the intervention group.
  Arms: Cold Debriefing
Behavioral: Hot Debriefing — The control group received a hot debriefing (immediately after the simulation).
  Arms: Hot Debriefing

SUMMARY:
The goal of this clinical trial is to find out if immediate (hot) or delayed (cold) debriefing is better for undergraduate nursing students during Basic Life Support (BLS) training.

The study aims to:

* Identify the effect of hot versus cold debriefing in BLS training for nursing students.
* Identify which debriefing method students prefer.

Researchers will compare the two debriefing methods. Participants will:

* Be randomly assigned (by flipping a coin) to either hot or cold debriefing.
* Take part in a simulation about Basic Life Support.

DETAILED DESCRIPTION:
This RCT aimed to identify the efficacy of cold versus hot debriefing in BLS training for undergraduate nursing students' BLS competence and to assess the impact of hot and cold debriefing nursing students' debriefing experience.

Specific Aims/Hypothesis Specific aim 1: Identify the efficacy of cold versus hot debriefing in BLS training for undergraduate nursing students' BLS competence.

Hypothesis 1a: In both cold and hot debriefing groups, there is a significant difference in the BLS competence of undergraduate nursing students between pre-intervention and post-intervention.

Hypothesis 1b: Undergraduate nursing students who receive cold debriefing will show greater BLS competence than those who receive hot debriefing. Our approach to testing the aim is to conduct an experimental design study.

Specific aim 2: Assess the impact of hot and cold debriefing on undergraduate nursing students' debriefing experience.

Hypothesis 2: Undergraduate nursing students who receive cold debriefing will show greater debriefing experience scores than those who receive hot debriefing.

ELIGIBILITY:
Inclusion Criteria:

* Junior or senior nursing students (i.e., in their third or fourth year of the BSN degree).

Exclusion Criteria:

* Nursing students who are not junior or senior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alanezi, PhD Candidate, MSc, BSN, Principal Investigator — University of Cincinnati
Locations (1):
- University Of Cincinnati College of Nursing, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Unending

REFERENCES:
- [Background] Kolb, D. A. (2014). Experiential learning: Experience as the source of learning and development (2nd ed.). Pearson Education, Inc.
- [Result] Reed, S. J. (2012). Debriefing experience scale: Development of a tool to evaluate the student learning experience in debriefing. Clinical Simulation in Nursing, 8(6), e211-e217.
- [Result] Meguerdichian M, Bajaj K, Ivanhoe R, Lin Y, Sloma A, de Roche A, Altonen B, Bentley S, Cheng A, Walker K. Impact of the PEARLS Healthcare Debriefing cognitive aid on facilitator cognitive load, workload, and debriefing quality: a pilot study. Adv Simul (Lond). 2022 Dec 12;7(1):40. doi: 10.1186/s41077-022-00236-x. PMID 36503623
- [Result] Ha EH. Effects of hot and cold debriefing in simulation with case-based learning. Jpn J Nurs Sci. 2021 Feb 26:e12410. doi: 10.1111/jjns.12410. Online ahead of print. PMID 33634592
- [Result] Kessler DO, Cheng A, Mullan PC. Debriefing in the emergency department after clinical events: a practical guide. Ann Emerg Med. 2015 Jun;65(6):690-8. doi: 10.1016/j.annemergmed.2014.10.019. Epub 2014 Nov 15. PMID 25455910
- [Result] Couper K, Perkins GD. Debriefing after resuscitation. Curr Opin Crit Care. 2013 Jun;19(3):188-94. doi: 10.1097/MCC.0b013e32835f58aa. PMID 23426138

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Debriefing | Hot Debriefing
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Debriefing | Hot Debriefing | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Finished Credits Hours in Current Program [Mean (Standard Deviation); unit: Credits Hours] | 92.6 (19.2) | 98.1 (17.7) | 95.3 (18.5)
Overall GPA [Mean (Standard Deviation); unit: GPA] | 3.62 (0.31) | 3.60 (0.29) | 3.61 (0.30)
BLS Certificate [Count of Participants; unit: Participants]
  Yes | 22 | 22 | 44
  No | 0 | 0 | 0
BLS Certificate Date [Count of Participants; unit: Participants]
  1 to 3 months | 7 | 7 | 14
  4 to 6 months | 5 | 6 | 11
  7 to 12 months | 4 | 2 | 6
  >1 year | 5 | 8 | 13
Simulation Experiences [Count of Participants; unit: Participants]
  Yes | 18 | 20 | 38
  No | 4 | 2 | 6
Simulation sessions [Count of Participants; unit: Participants]
  None | 4 | 2 | 6
  1-3 | 14 | 17 | 31
  4-6 | 2 | 2 | 4
  >6 | 2 | 1 | 3
Previous cardiac arrest(s) [Count of Participants; unit: Participants]
  None | 15 | 15 | 30
  1-3 | 5 | 4 | 9
  4-6 | 2 | 2 | 4
  >6 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Basic Life Support Competence
Description: Competence level was measured via the American Heart Association (2020) Basic Life Support competency checklist, which is a dichotomous rating scale of 0 (not done/done incorrectly) and 1 (done correctly); there was a total of 15 points. The higher the score, the better the outcome.
Time Frame: Immediately after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cold Debriefing | Hot Debriefing
Number analyzed (Participants) | 22 | 22
score on a scale
  Baseline Score | 9.45 (2.93) | 10.04 (1.70)
  Post-test Score | 14.63 (5.18) | 14.54 (4.5)
Statistical Analysis 1: Comparison: Cold Debriefing vs Hot Debriefing; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.09

2. Secondary Outcome: Debriefing Experience Scale
Description: The Debriefing Experience Scale (DES) (Reed, 2012) was developed to assess nursing students debriefing experience. It included 20 elements in total and was split into four subscales: (1) Analyzing Thoughts and Feelings; (2) Learning and Makin Connections; (3) Facilitator Skill in Conducting the Debriefing; and (4) Appropriate Facilitator Guidance (Reed, 2012). A Likert scale ranges from 1 (strongly disagree) to 5 (strongly agree). The minimum score is 20 and the maximum is 100. The higher the score, the better the outcome.
Time Frame: Immediately after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cold Debriefing | Hot Debriefing
Number analyzed (Participants) | 22 | 22
score on a scale
  Total Opinion | 95.68 (6.06) | 93.63 (8.06)
  Total Importance | 93.86 (7.21) | 92.18 (9.84)

ADVERSE EVENTS:
Time Frame: The study did not collect data on adverse events. It was a simulation experience where we tested two debriefing methods and their impact on BLS competence for undergraduate nursing students.
Arm/Group | Cold Debriefing | Hot Debriefing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We initially aimed to recruit 52 participants but ended up with only 44. This may pose a threat to the internal validity of the study. Additionally, since the participants were drawn from a single nursing school, the generalizability of the findings is limited, representing a threat to external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06624449/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06624449/SAP_001.pdf